CLINICAL TRIAL: NCT03869411
Title: Effects of Exercise Intervention and Confounding Factors on Type II Diabetic Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201812135RINB
Record Dates: First submitted 2019-03-05; First posted 2019-03-11 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Diabetes and Healthy Control; FTO Gene Expression; Aerobic Exercise Intervention or Home Exercise; Pre-training and Post-training
Keywords: diabetes; muscle quality; aerobic exercise; FTO gene
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: his study is going to recruit subjects with and without type 2 diabetes and age between 30 and 70 years old. This study will be focused on the effects of diabetes on maximum aerobic exercise intensity (VO2max) and muscle quality including microcirculation (by NIRS), mechanical properties (by elastography) and isometric strength in different age groups, and observe whether these results are related to the clinically relevant findings of diabetes. This study will recruit qualified diabetic subjects according to their results of maximal aerobic exercise capacity (VO2max) and assign them into two groups; aerobic exercise or home exercise intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aerobic exercise group (Experimental): This study will recruit qualified diabetic subjects according to their results of maximal aerobic exercise capacity (VO2max) and assign them into aerobic exercise or home exercise groups, based on their willingness. The aerobic exercise group will arranged to the supervised aerobic dance program, it's consisted of 50 mins per session, 3 sessions per week and last for 3 months.
  Interventions: Behavioral: supervised aerobic exercise or home-based aerobic exercise
- home exercise group (Experimental): This study will recruit qualified diabetic subjects according to their results of maximal aerobic exercise capacity (VO2max) and assign them into aerobic exercise or home exercise groups, based on their willingness.The home exercise group will give the exercise recommendation based on ACSM's guideline, and it's consisted of 50 mins per session, 3 sessions per week and last for 3 months.
  Interventions: Behavioral: supervised aerobic exercise or home-based aerobic exercise
- health control group (Active Comparator): This study will recruit subjects without type 2 diabetes and the age matched to the diabetes groups.
  Interventions: Behavioral: supervised aerobic exercise or home-based aerobic exercise

INTERVENTIONS:
Behavioral: supervised aerobic exercise or home-based aerobic exercise — The aerobic exercise and home exercise programs are consisted of 50 minutes per time, 3 times per weeks and totally 3 months.
  The aerobic exercise group will perform the exercise program under one physical therapy and one aerobic dance teacher supervised. The home exercise group will do the exercise program based on ACSM's aerobic exercise recommend, and will used the home exercise record form to make sure their cooperation.

SUMMARY:
The aim of the first year of this three-year plan is to analyze and compare the muscle quality of lower limb muscle (microcirculation, muscle performance and mechanical characteristics) and maximal aerobic exercise capacity in treadmill exercise tests for diabetic and non-diabetic cases. The hypotheses are:1) the muscle quality of lower limb muscle and maximal aerobic exercise capacity are different between participate with diabetic and non-diabetic, 2) the effect of the three-month aerobic exercise intervention or home exercise on the characteristics of the muscle quality are different , and 3) intrinsic factors (such as age, BMI, and HDL) and characteristics of specific FTO genes are influenced the training outcomes.

DETAILED DESCRIPTION:
Participants with diabetes will attend an 12-week aerobic exercise intervention or home exercise if the exercise test result of the maximum rate of oxygen consumption is fair or poor. Assessments will be taken before and after the training program, which including muscle strength, stiffness, quality, microcirculation and exercise capacity. Comparisons between the pre-training and post-training condition will be made for each groups. And the assessments also compare with the healthy control group.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes group: 1) Age between 30-70 years of old, 2) type 2 diabetes.
* Healthy control group: 1) Age between 30-70 years of old, 2) without diabetes

Exclusion Criteria:

* history of moderate-severe somatic or autonomic neuropathy, cardiovascular disease, preproliferative or proliferative retinopathy, and chronic renal failure
* unable to perform the programs or assessments
* other systematic diseases

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
index of muscle stiffness | Change from Baseline muscle quality at 3 months
  elastography was used, units on kPa
muscle strength of knee extensor and plantarflexor | Change from Baseline functional performance at 3 months
  Dynamometer was used to measure muscle strength, units on kilograms
Relative sliding of muscles | Change from Baseline muscle quality at 3 months
  B mode sonography was used, units on mm/s
muscle microcirculation | Change from Baseline muscle quality at 3 months
  Near-infrared spectroscopy was used to measure oxygen saturation on muscle, units on percentage
maximum rate of oxygen consumption | Baseline
  Bruce treadmill protocol was used in the maximal exercise testing, maximum rate of oxygen consumption record as ml/kg/min

SECONDARY OUTCOMES:
characteristics of specific FTO genes | Baseline
  rs9939609 SNP analysis, record as TT or TA or AA type
physical activity level | Change from Baseline functional performance at 3 months
  self report the ability of walking one-fourth of a mile, record as degree of difficulty: none, some difficulty, much difficulty, inability
BMI | Change from Baseline functional performance at 3 months
  weight and height will be combined to report BMI in kg/m^2
blood glucose level | Change from Baseline functional performance at 3 months
  Hemoglobin A1c (HbA1c), unit on percentage
blood cholesterol | Change from Baseline functional performance at 3 months
  total cholesterol, units on mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Colberg SR, Sigal RJ, Fernhall B, Regensteiner JG, Blissmer BJ, Rubin RR, Chasan-Taber L, Albright AL, Braun B; American College of Sports Medicine; American Diabetes Association. Exercise and type 2 diabetes: the American College of Sports Medicine and the American Diabetes Association: joint position statement executive summary. Diabetes Care. 2010 Dec;33(12):2692-6. doi: 10.2337/dc10-1548. No abstract available. PMID 21115771
- [Result] Bacchi E, Negri C, Zanolin ME, Milanese C, Faccioli N, Trombetta M, Zoppini G, Cevese A, Bonadonna RC, Schena F, Bonora E, Lanza M, Moghetti P. Metabolic effects of aerobic training and resistance training in type 2 diabetic subjects: a randomized controlled trial (the RAED2 study). Diabetes Care. 2012 Apr;35(4):676-82. doi: 10.2337/dc11-1655. Epub 2012 Feb 16. PMID 22344613
- [Result] Prior SJ, Blumenthal JB, Katzel LI, Goldberg AP, Ryan AS. Increased skeletal muscle capillarization after aerobic exercise training and weight loss improves insulin sensitivity in adults with IGT. Diabetes Care. 2014 May;37(5):1469-75. doi: 10.2337/dc13-2358. Epub 2014 Mar 4. PMID 24595633